CLINICAL TRIAL: NCT03677414
Title: Analysis of Androgene Receptors Axis and DNA Damage Repair Genes From Plasma DNA (ctDNA) in Patients With Prostate Cancer
Brief Title: Analysis of Androgene Receptors Axis and DNA Damage Repair Genes in Patients With Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: FWF Project KLI 710-B26; 21-228 ex 09/10 (Other: Ethics Committee at Med Uni Graz)
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Prostatic Neoplasms
Keywords: circulating-tumor DNA ctDNA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma DNA Primary tumor Buccal swap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this project, we would like to focus on castration-sensitive prostate cancer (CRPC). This is a highly variable clinical picture with differentiated and burdening symptoms. The clinical parameters used to estimate the prognosis have so far only shown a very limited valence; genetic markers have so far only rarely been investigated.

In the course of our preliminary investigations, we were already able to isolate 189 plasma samples from 59 patients with metastatic prostate cancer. These samples are prepared by highly innovative techniques, e.g. "whole genome sequencing", in order to gain comprehensive insights into the spectrum of genetic changes under therapy and the associated tumor evolution. These results should be compared with the genetic material of the respective prostate tumors, which originate from previous operations. This highly comprehensive data, which will yield results on copy number changes, mutations, and gene expression, will allow analysis of signaling pathways of unprecedented resolution to increase the efficacy of targeted therapies in patients and minimize the burden of non-effective therapy side effects.

DETAILED DESCRIPTION:
The investigators collected 189 plasma samples from 59 patients with metastasized CRPC treated with abiraterone/enzalutamide. In order to stratify plasma DNA samples based on the presence of low (i.e. z-score ≤5; corresponds to <10% ctDNA) versus high (z-score >5; corresponds to ≥10% ctDNA) genomic complexity in ctDNA the investigators employed the modified Fast Aneuploidy Screening Test-Sequencing System (mFAST-SeqS), which provides a plasma based marker of aneuploidy (z-score). Altogether 106 plasma samples with a low z-score will be evaluated only with the AVENIO ctDNA Expanded Kit, which is capable of detecting mutations with VAFs as low as 0.1% . From the 83 plasma samples with increased z-score will be sequenced with high coverage (70x) so that both mutations and nucleosome positions can be extracted from the obtained sequences. With the other 32 high z-score samples plasma-Seq will be conducted to establish genome-wide copy number profiles and 31 prostate cancer genes will be enriched to screen for mutations in these genes.

At present, there is no evidence what parameters should be used to decide which treatment options are best for metastatic prostate cancer patients. The suggested innovative technologies, i.e. nucleosome position mapping and gene expression analyses will provide systematic maps of nucleosome positions. The sequencing of plasma samples with 70x will provide in addition a comprehensive view on the mutation spectrum in metastatic prostate cancer. By inclusion of primary tumor analyses, an unprecedented view on prostate cancer genome Evolution will be obtained. Overall, the comprehensive data set (copy number changes, mutations, gene expression) will allow pathway analyses with unprecedented resolution.

ELIGIBILITY:
Inclusion Criteria:

* subject has proven histological diagnosis of prostate cancer
* subject was treated with abiraterone and/or enzalutamide.

Exclusion Criteria:

* patient rejects the participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes men with metastasized prostate cancer.
Study Population: The study includes men with proven histological diagnosis of prostate cancer and treatment with abiraterone and/or enzalutamide.
  Participants were recruited at the Medical University Hospital of Graz.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Nucleosome positioning patterns | 3 years
  Here, samples with increased z-score (z-score >5; corresponds to ≥10% ctDNA; modified Fast Aneuploidy Screening Test-Sequencing System (mFAST-SeqS)) will be sequenced with high coverage (70x) so that nucleosome positions can be extracted from the obtained sequences. As at TSSs (transcriptional start site), the nucleosome occupancy results in different read-depth coverage patterns in expressed and silent genes (Ulz et al., Nat Genet 2016), systematic maps of nucleosome positions in defined patients will be generated.

SECONDARY OUTCOMES:
Focal amplifications in ctDNA | 3 years
  Mapping (absolute number and size) of recurrent focal amplifications/gained regions and identification of the driver genes within these amplicons by systematic cataloging of genes expressed in focal amplifications/gained regions. In order to facilitate the identification of focal amplifications we apply very stringent/conservative criteria regarding amplicon size and gene density, which we applied in previous publications (Ulz et al., Nat Commun 2016; Ulz, Heitzer, Speicher, Nat Genet 2016).
Prostate Cancer Panel | 3 years
  Characterization of mutation frequency of enriched prostate cancer genes using plasma-Seq (i.e. AKAP9, APC, AR, ATM, BRAF, BRCA1, BRCA2, CTNNB1, EGFR, ERG, FOXA1, GNAS, GRIN2A, HRAS, KRAS, MED12, MLL, MLL2, MLL3, MLLT3, NOTCH1, NRG1, PIK3CA, PIK3CB, PIK3R1, PTEN, RB1, SPOP, TMPRSS2, TP53, ZFHX3).
Clinico-pathological characteristics | 3 years
  Documentation of clinico-pathological characteristics (PSA, NSE; blood count; localization, number and size of metastases by imaging) including prior and subsequent therapies.To identify predictive/prognostic biomarkers, newly occurring genomic changes in the plasma DNA (see primary outcome and further secondary outcome measures) will be correlated with outcomes of given therapies.
Analyses of primary tumors | 3 years
  Measurement of copy number changes in primary tumors by next-generation sequencing, i.e. SCNA-seq, and RNA-Seq for comparison with the nucleosome positions, see above.
Buccal swap | 3 years
  Distinction germ line vs. somatic mutations

CONTACTS AND LOCATIONS:
Overall Officials: Jochen B Geigl, Prof, MD, Principal Investigator — Institute of Human Genetics
Locations (1):
- Institute of Human Genetics, Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Ulz P, Belic J, Graf R, Auer M, Lafer I, Fischereder K, Webersinke G, Pummer K, Augustin H, Pichler M, Hoefler G, Bauernhofer T, Geigl JB, Heitzer E, Speicher MR. Whole-genome plasma sequencing reveals focal amplifications as a driving force in metastatic prostate cancer. Nat Commun. 2016 Jun 22;7:12008. doi: 10.1038/ncomms12008. PMID 27328849
- [Background] Ulz P, Heitzer E, Speicher MR. Co-occurrence of MYC amplification and TP53 mutations in human cancer. Nat Genet. 2016 Feb;48(2):104-6. doi: 10.1038/ng.3468. No abstract available. PMID 26813759
- [Background] Ulz P, Thallinger GG, Auer M, Graf R, Kashofer K, Jahn SW, Abete L, Pristauz G, Petru E, Geigl JB, Heitzer E, Speicher MR. Inferring expressed genes by whole-genome sequencing of plasma DNA. Nat Genet. 2016 Oct;48(10):1273-8. doi: 10.1038/ng.3648. Epub 2016 Aug 29. PMID 27571261
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306